CLINICAL TRIAL: NCT06913530
Title: European Multicentre Study of Long-term Results Following Visceral Arteries Revascularization: the E-VisAR Study
Acronym: E-VisAR
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Nicola Leone, Principal Investigator, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: E-VisAR
Record Dates: First submitted 2025-02-13; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Visceral Artery Aneurysm; Mesenteric Artery Ischemia; Renal Artery Aneurysm; Renal Artery Stenosis; Renal Artery Stenosis Atherosclerotic; Renal Artery Fibromuscular Dysplasia; Chronic Mesenteric Ischemia; Visceral Artery Dissection; Mesenteric Artery Dissection
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective patients: Patients who have undergone visceral vessels revascularization of any kind up to 20 years prior to the study launch.
- Prospective patients: Patients enrolled in the study for a visceral vessel revascularization of any kind after the study launch.

SUMMARY:
Visceral arteries pathologies are a broad-spectrum of conditions with an extremely low incidence, estimated at 9.2% and 6.2% per 100,000 inhabitants for chronic and acute mesenteric ischemia, respectively, and 0.01-0.2% for aneurysms. The literature regarding the topic is limited in number and fragmented, having multiple vessels involved along with rare conditions caused by different aetiologies. However, these diseases are of utmost importance considering that acute presentation is common and the treatment in urgent setting is challenging and still facing high mortality rates. There are still several grey areas regarding the treatment of these pathologies. The last decades showed an increasing utilization of an endovascular approach to treat visceral vessel diseases. On one hand, the early- and mid-term superiority of endovascular revascularization vs. open surgical repair has been demonstrated considering the reduction of morbidity and mortality, and length of stay. However, publications reporting long-term (> five years) are still lacking.

This study is a real-word, ambispective, multi-arm, multicenter study that aims to evaluate the long-term results of visceral vessel revascularization in different diseases, districts, and approaches. Patients will be divided according to the target vessel and index disease. For each subgroup, a comparison between endovascular and open repair will be performed.

The primary outcome is to compare endovascular and open approach in terms of survival, further divided into overall and disease-related mortality, during long term follow-up (> 5 years). Moreover, early and mid-term data should be considered to provide reliable results. This outcome will be stratified as well within each disease- specific arm.

At the study launch, data collection of patients who have undergone visceral vessels revascularization in the previous 20 years will begin. At the same time, all new cases of visceral vessel revascularization will be proposed for enrollment and follow-up in the prospective arm. The retrospective cohort will provide informative results regarding the long-term survival of these patients. This information will be used to adjust the sample size for the prospective cohort.

DETAILED DESCRIPTION:
The 'European Multicentre Study of Long-term Results Following Visceral Arteries Revascularization: the E-VisAR study' is a real-word, ambispective, multi-arm, multicenter study that aims to evaluate the long-term results of visceral vessel revascularization in different diseases, districts, and approaches. Patients will be divided according to the target vessel and index disease. For each subgroup, a comparison between endovascular and open repair will be performed.

Given the study design and the current state of knowledge, here are some potential expected results:

Long-Term Survival Comparison:

The primary expectation is to provide robust, long-term data comparing endovascular and open surgical repair in visceral artery revascularization.

It's possible that the study will confirm the early and mid-term benefits of endovascular procedures in terms of reduced morbidity and mortality, extending these findings to long-term outcomes. However, it's also possible that certain subgroups (e.g., specific diseases, specific vessel involvement) may show different long-term results, with open repair potentially demonstrating superiority in some cases. Endovascular approach may demonstrate higher rate of re-intervention, or lower long term patency for certain diseases.

Disease-Specific Outcomes:

The study will likely reveal variations in outcomes based on the specific disease (e.g., chronic mesenteric ischemia vs. aneurysms). For example, aneurysms might show different long-term patency rates compared to stenotic lesions.

Identification of Risk Factors:

The large dataset will allow for the identification of risk factors associated with adverse long-term outcomes, such as specific comorbidities, anatomical variations, or procedural factors.

Refinement of Treatment Guidelines:

The long-term data will contribute to refining treatment guidelines for visceral artery pathologies, helping to optimize patient selection and procedural techniques.

Real World data:

This study will provide real world data, which is very important to validate the results of randomized control trials, which are often conducted on selected populations. In addition, randomized control trials have not been performed in this field and will likely never happen looking at the diseases limitations.

Relevance for Patients:

Improved Treatment Decisions:

Patients will benefit from more informed treatment decisions, as the study will provide clearer evidence on the long-term effectiveness of different revascularization approaches. This will lead to more personalized treatment plans, tailored to individual patient needs and risk factors.

Reduced Morbidity and Mortality:

By identifying optimal treatment strategies, the study has the potential to reduce morbidity and mortality associated with visceral artery pathologies.

Improved Quality of Life:

Successful revascularization can alleviate symptoms, improve nutritional status, and enhance the overall quality of life for patients with these conditions.

Better understanding of rare diseases:

These diseases are rare, and this study will provide more information to patients that suffer from them.

Relevance for Physicians:

Evidence-Based Practice:

The study will provide valuable evidence to support clinical decision-making, moving away from anecdotal experience and towards evidence-based practice.

Refined Treatment Strategies:

Physicians will gain a better understanding of the long-term outcomes of different revascularization techniques, allowing for more precise and effective treatment strategies.

Identification of High-Risk Patients:

The study will help identify patients at high risk for adverse outcomes, enabling physicians to implement preventive measures and closer monitoring.

Improved Patient Selection:

The data will help physicians to select the best treatment approach for each individual patient.

Contribution to the Field:

The study will contribute to the advancement of knowledge in the field of visceral artery pathologies, ultimately leading to better patient care.

Due to the multicenter nature of the study, this will help to standardize the care of these rare pathologies. In essence, the study is crucial for filling the knowledge gap regarding the long-term outcomes of visceral artery revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with atherosclerotic disease, aneurysms, or dissection;
* Pathologies involving one or more visceral vessels (celiac, mesenteric, renal arteries, and their branches);
* Patients receiving revascularization, both surgical and endovascular, in elective and urgent/emergent settings;
* For the retrospective cohort, patients who underwent revascularization up to 20 years from the study launch regardless of the follow-up time.

Exclusion Criteria:

* Absence of follow-up imaging available and/or reported in follow-up medical reports;
* For the retrospective cohort, a follow-up shorter than three years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Starting from the study launch, all patients with indication for visceral vessel revascularization will be referred to the study staff for enrollment in the prospective cohort. Assessment of the patient will be performed by a vascular surgeon being part of the Medical Staff. After revascularization, clinical and imaging outcomes will be evaluated at short- (within one year), mid- (three-five years), and long-term (> five years) follow-up.
  For the retrospective cohort, patients' enrollment eligibility (inclusion/exclusion criteria are listed below) and anamnestic, clinical, and morphological data will be reviewed and collected. Data collection for the retrospective cohort will include all eligible patients who have undergone visceral vessels revascularization up to 20 years from the study launch and regardless of the follow-up time.
  The two cohorts will be independently followed during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | one, three, and five years
  The primary outcome is to compare endovascular and open approach in terms of survival, further divided into overall and disease-related mortality. The outcome will be evaluated at early, mid-, and long-term follow-up, one, three, and five years respectively. This outcome will be stratified as well within each disease- specific arm.

SECONDARY OUTCOMES:
Technical success | one, three, and five years
  defined as successful revascularization meaning correct device positioning with <30% residual stenosis in case of stenotic/occlusive disease, correct sealing without endoleak in case of aneurysm exclusion, or the abscence of reperfusion for coils embolization of aneurysmal disease. The success is given without technical issue hindering device positioning and with no complication occurring during the intervention.
Clinical success | one, three, and five years
  To compare endovascular and open approach in term of early, mid-, and long-term clinical success, meaning the absence of specific symptoms recurrence and revascularized vessel patency or successful aneurysm exclusion without endoleaks or reperfusion and aneurysm growth following embolization.
Long-term patency | one, three, and five years
  To compare endovascular and open approaches in terms of early, mid-, and long-term patency, divided into primary, secondary, and assisted patency. Primary patency will be given if the revascularized artery will be patent at the time point. Secondary patency will be given for the patent artery following a reintervention performed for occlusion. Assisted patency will be given for those arteries requiring additional, non-planned, intervention aimed at maintaining patency, e.g. in case of severe stenosis.
Reintervention rates | one, three, and five years
  To compare endovascular and open approach in term of long term reintervention rates, divided those performed for endoleak, aneurysm growth, restenosis, and occlusion based on index treatment.